CLINICAL TRIAL: NCT04486144
Title: Impact of a Proprietary Extract of Nerium Oleander on Immune Function as Evidenced by Clinical Symptoms and Mortality :A Feasibility Study
Brief Title: Impact Nerium Oleander on Immune Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthQuilt (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 052020
Record Dates: First submitted 2020-07-20; First posted 2020-07-24 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Covid19 Positive Patient; Covid19 Close Contact; Immune Function
Keywords: Covid19; Nerium oleander; Clinical symptoms; Mortality; Immune Function
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- COVID19 Positive: Intervention Group (Receive extract) (Experimental): These are patients that are COVID19 positive who elect to try the extract.
  Interventions: Other: Proprietary extract of Nerium oleander
- COVID19 Positive: Comparison Group (Do NOT receive extract) (No Intervention): These are patients that are COVID19 positive who do NOT elect to try the extract
- COVID19 Exposed: Intervention Group (Receive extract) (Experimental): These are patients that are COVID19 negative at the start, live with a COVID19 positive patient and who elect to try the extract.
  Interventions: Other: Proprietary extract of Nerium oleander
- COVID19 Exposed: Comparison Group (Do NOT receive extract) (No Intervention): These are patients that are COVID19 negative at the start, live with a COVID19 positive patient and who elect to NOT try the extract.

INTERVENTIONS:
Other: Proprietary extract of Nerium oleander — This is a proprietary extract of Nerium oleander that is 6.25 ug per 0.5 ml of suspension. It is administered sublingually every six hours for 5 days. The daily dose is 25 ug and the 5 day dose is 125 ug.
  Arms: COVID19 Exposed: Intervention Group (Receive extract); COVID19 Positive: Intervention Group (Receive extract)

SUMMARY:
Assess the impact of a proprietary extract of Nerium oleander on immune function as evidenced by COVID-19 symptoms and mortality in COVID-19 positive patients and their close contacts compared to controls that did not receive the extract.

DETAILED DESCRIPTION:
This is an exploratory study based on positive in-vitro, and in-vivo (humans) that appear to support an immune function benefit. Up to 100 patients that are COVID-19 positive in the ambulatory setting will be invited to participate. After informed consent is obtained, patients will be in either the Intervention Group (receive extract) or Comparison Group (did not receive extract). A baseline assessment and record review will be conducted to assure eligibility criteria. Patients in the Intervention Group will be given .5 ml (6.25 mg of extract) every 6 hours for 5 days, total of 25 mg per day / 125 mg for 5 days. Patient vital signs (temperature, pulse oximetry, blood pressure) and CDC symptoms / side effects will also be tracked. A dedicated medical oversight team with 24 / 7 access to care will be provided to monitor safety and tolerance. Patients will be followed for 10 days. Baseline antibody, RT-PCR, and live virus will be collected on Day 1, Day 5, and Day 10. A Data Monitoring Committee at the Schull Institute will meet weekly to review data.

ELIGIBILITY:
Inclusion Criteria:

* Age 18
* COVID 19 positive or close contact of COVID 19 positive
* No use of cardiac glycosides or other antiarrhythmic medications

Exclusion Criteria:

* No use of cardiac glycosides or other antiarrhythmic medications
* No allergy to coconut oil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2020-07-23 (Actual)

PRIMARY OUTCOMES:
COVID19 symptoms | Every 6 hours for 10 days
  The CDC list of symptoms and "other".
Mortality | 10 days from enrollment into the Study, e.g. Day 10
  A patient in any arm that dies.

SECONDARY OUTCOMES:
COVID19 Live Virus | Day 1, Day 5, Day 10
  COVID19 Live Virus Nasopharyngeal swab performed by UTMB, Texas
RT-PCR COVID19 Test | Day 1, Day 5, Day 10
  RT-PCR Nasopharyngeal swab performed by Fulgent, California

CONTACTS AND LOCATIONS:
Overall Officials: Kim Dunn, MD, Ph.D., Principal Investigator — KDunn and Associates, PA dba Healthquilt
Locations (1):
- KDunn and Associates, PA, dba Healthquilt, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
KDunn and Associates, PA will de-identify data and archive it at The Schull Institute Data Archive at the University of Texas School of Biomedical Informatics after the Summer Research Program Conclusion.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: October 2020
Access Criteria: Need to have a specific question or plan to study further.
URL: http://www.theschullinstitute.org

REFERENCES:
- See also: Plante KS, Plante JA, Fernandez D, et al. Prophylactic and therapeutic inhibition of in vitro SARS-CoV-2 replication by Oleandrin. bioRxiv. July 15, 2020. Cold Spring Harbor Laboratory. — http://doi.org/10.1101/2020.07.15.203489